CLINICAL TRIAL: NCT04933006
Title: Hemodialysis-Induced Blood Pressure Change As A Prognostic Factor In End-Stage Renal Disease
Brief Title: Hemodialysis-Induced Blood Pressure Change In End-Stage Renal Disease
Acronym: Hemodialysis
Status: Completed | Type: Observational
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Director, Shahid Beheshti University of Medical Sciences
Other Study IDs: SBMU326
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Hemodialysis
Keywords: Echocardiography
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pulsevelocity — arterial stiffness evaluation with pulsewave velocity
  Other Names: Echocardiography

SUMMARY:
Cardiovascular events are still the leading cause of mortality and morbidity in patients with ESRD including hemodialysis patients . Although the conventional risk factors of CVD are relatively recognized in general population, an inverse epidemiologic relationship has been reported for many CV risk factors in CKD patients, including hypertension, BMI and lipid profile .Therefore, a comprehensive investigation is necessary to be able to do effective risk management strategies in this population and some surrogate markers are required to be determined for illustrating the net effect of the risk factors.

While several mechanisms have been attributed to hypertension in hemodialysis (HD) patients, the exact pathogenesis, impact, monitoring and control of hypertension in HD patients are still challenging subjects in clinical nephrology. Both low and high BP associate with higher mortality in HD. But a reliable marker for defining an optimal BP in HD is still an important question.

It seems that arterial stiffness play an axial role in the cardiovascular and renal adverse outcomes in CKD and HD, as it is in several other populations , Arterial stiffness has been demonstrated as an independent predictor of mortality in hemodialysis patients . However, hemodialysis patients experience a fluctuating hemodynamic state and there are several limitations for consecutive measurement of arterial stiffness indices such as pulse wave velocity (PWV). Furthermore, the expensive measurement devices and expert operators might not be available in every dialysis center.

DETAILED DESCRIPTION:
From 60 patients who were on a HD program in a HD center in a referral hospital, fifty one individuals were included into the study. Patients on maintenance hemodialysis, for at least 12 hours per weeks were included into the study. But, patients with symptomatic CVD, AV fistula on both arms, acute deteriorating states and any recent major trauma or patients who refused measurements were excluded. No change in their current medication was administered. All patients were on maintenance HD for at least 12 months and were assumed as good volume controlled. Dialysis protocol with a mean sp KT/V = 1.4/ session, using Bicarbonate dialysate, dialysate flow rate = 500cc /min was applied by Fresenius B 4008machine. BP was measured using a validated automated device (Omron-HBP1300). Pulse wave analysis was performed using the SphygmoCor (Sydney, Atcor Medical®,2005) to assess Augmentation Index (AIx) as a surrogate for arterial stiffness, as well as several hemodynamic measures at the recruitment and repeated in alive individuals after 5 years of follow-up. Similarly Echocardiography was employed at the beginnings and repeated at the end of the study by EKO 7 Cardiovascular Ultrasound System (Samsung Medison©). A single observerwas responsible for each series of measurements, double checked.

ELIGIBILITY:
Inclusion Criteria:

* Patients on maintenance hemodialysis for at least 12 hours per weeks

Exclusion Criteria:

* Patients with symptomatic CVD
* Recent major trauma
* Patients who refused measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on maintenance hemodialysis, for at least 12 hours per weeks were included into the study. But, patients with symptomatic CVD, AV fistula on both arms, acute deteriorating states and any recent major trauma or patients who refused measurements were excluded. No change in their current medication was administered. All patients were on maintenance HD for at least 12 months and were assumed as good volume controlled.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
mortality | during the six month post starting hemodialysis
  percentage of mortality during hemodialysis due to blood pressure changes

CONTACTS AND LOCATIONS:
Overall Officials: SBMU SBMU, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- SBMU, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No